CLINICAL TRIAL: NCT04583007
Title: Expanded Access Program: Lanadelumab for the Prevention of Acute Attacks of Hereditary Angioedema (HAE) in Pediatric Patients 2 to <12 Years of Age and Lanadelumab for the Prevention Against Acute Attacks of Non-histaminergic Angioedema With Normal C1-Inhibitor (C1-INH)
Brief Title: Expanded Access for the Prevention of Acute Attacks of 1) Hereditary Angioedema (HAE) in Children and 2) Non-histaminergic Angioedema With Normal C1-Inhibitor (C1-INH) in Teenagers and Adults
Status: No longer available | Type: Expanded Access
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: TAK-743-6001; TAK-743-5012 (Other: Takeda)
Record Dates: First submitted 2020-10-01; First posted 2020-10-12 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Hereditary Angioedema (HAE); Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema | interventions — lanadelumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Lanadelumab 150 mg — TAK-743-6001: Participants will receive subcutaneous (SC) injection of lanadelumab at a dose of 150 milligrams (mg) at the same frequency (for every 2 weeks [Q2W] or for every 4 weeks [Q4W]) given at the completion of SPRING study until benefit-risk no longer favors the individual participant or an appropriate alternative therapy becomes available or lanadelumab 150 mg/ 1 milliliter (mL) becomes commercially available or the participants turns 12 years of age or participant chooses to discontinue treatment. For participants aged 6-12 years, a dose frequency may be modified based on a benefit-risk assessment and medical decision from the treating physician.
  Other Names: TAK-743; SHP643; DX-2930
Drug: Lanadelumab 300 mg — TAK-743-5012: Participants will receive SC injection of lanadelumab in prefilled syringe at a dose of 300 mg, Q2W or Q4W if well controlled for 26 weeks across Study TAK-743-3001 and this (TAK-743-5012) program.
  Other Names: TAK-743; SHP643; DX-2930

SUMMARY:
The expanded access program allows people to gain access to an unlicensed treatment on compassionate grounds. Lanadelumab, also known as TAK-743, is a medicine to help prevent angioedema attacks. This expanded access program enables these participants with a high unmet medical need to continue receiving lanadelumab during the interim period between completion of either the SHP643-301 (NCT04070326; SPRING study) or the TAK-743-3001 (NCT04444895) study and potential licensure of lanadelumab for the respective age group and/or treatment.

ELIGIBILITY:
Inclusion Criteria:

TAK-743-6001 Study (Acute Attacks of HAE):

* Pediatric participants, 2 to <12 years of age, with HAE who completed the SHP643-301 (SPRING) study and are deriving continued clinical benefit from lanadelumab treatment will be invited to take part in this program
* Participants have no suitable alternative treatment options and cannot enter a lanadelumab clinical trial
* Participant has a parent(s)/legal guardian who is informed of the nature of the expanded access program and can provide written informed consent for the child to participate (with assent from child when appropriate) prior to treatment
* Participants does not have any of the following liver function test abnormalities : alanine aminotransferase (ALT) greater than (>)3x upper limit of normal (ULN), or aspartate aminotransferase (AST) >3x ULN, or total bilirubin >2x ULN (unless the bilirubin elevation is a result of Gilbert's syndrome)
* Participant does not have any condition that in the opinion of the Investigator may compromise their safety
* Participant does not have a known hypersensitivity to lanadelumab or its components
* Participant (greater than or equal to >or=6 years) and/or caregiver is willing to self-administer lanadelumab at home and has received documented training on self-administration during the SHP643-301 (SPRING) Study

For Female participants of childbearing potential only:

* Participant has agreed to be abstinent or agreed to comply with the applicable contraceptive requirements of this protocol for the duration of the expanded access program and for 70 days after completion
* Participant is not pregnant or breast-feeding Note: Participants who do not satisfy the above criteria will be excluded.

TAK-743-5012 Study (Acute Attacks of Non-histaminergic Angioedema With Normal C1-Inhibitor (C1-INH)):

* Participant has completed the treatment period of the TAK-743-3001 study (all Visit 14 assessments have been completed).
* Participant is demonstrating continued benefit from lanadelumab treatment.
* Participant and/or a parent(s)/legal guardian is informed of the nature of the expanded access program and can provide written informed consent for themselves or the child to participate (with assent from child when appropriate) prior to treatment).
* Participant does not have any condition including lab test that in the opinion of the Investigator may compromise their safety.
* Participant does not have a known hypersensitivity to lanadelumab or its components.
* Participant and/or caregiver is willing to self-administer lanadelumab at home and has received documented training on self-administration during the Study TAK-743-3001 OR the participant and/or caregiver is willing to self-administer lanadelumab at home and will receive training at the first two dose administrations in accordance with protocol.

Female Participants of childbearing potential only:

* Participant has agreed to be abstinent or agreed to comply with the applicable contraceptive requirements of this protocol for the duration of the expanded access program and for 70 days after completion of the last dose.
* Participant is not pregnant or breast-feeding.

Male Participants only:

* Participant has agreed to comply with the applicable contraceptive requirements of this protocol for the duration of the expanded access program and for 70 days following the last dose of lanadelumab
* Participant has agreed to not donate sperm during the course of the program and for 70 days following the last dose of lanadelumab.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (20):
- United States (14):
  - Medical Research of Arizona, Scottsdale, Arizona
  - AIRE Medical of Los Angeles, Santa Monica, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Henry J. Kanarek- Allergy, Asthma & Immunology, Overland Park, Kansas
  - Institute Asthma and Allergy, Chevy Chase, Maryland
  - Institute For Asthma and Allergy, Chevy Chase, Maryland
  - University of Michigan Allergy and Immunology Specialty Clinic, Ann Arbor, Michigan
  - Hudson-Essex Allergy, Belleville, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Clinical Research Center of Charlotte, Charlotte, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Toledo Institute of Clinical Research Asthma & Allergy Center, Toledo, Ohio
  - AARA Research Center, Dallas, Texas
- Yang Medicine, Ottawa, Ontario, Canada
- Germany (3):
  - Charité - Universitätsmedizin Berlin., Berlin
  - Klinikum der Johann-Wolfgang Goethe-Universitat., Frankfurt
  - Hämophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- Semmelweis Egyetem., Budapest, Hungary
- Hospital Universitario La Paz. Paseo de la Castellana, Madrid, Spain

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f9c5f412f8e61001ef32419?idFilter=%5B%22TAK-743-6001%22%5D